CLINICAL TRIAL: NCT06405412
Title: Effects of Malnutrition on Respiratory and Renal Functions in Patients Undergoing Peroral Endoscopic Myotomy (POEM)
Status: Recruiting | Type: Observational
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Zeliha Alicikus, Chief Anesthesiologist, Umraniye Education and Research Hospital
Other Study IDs: UERH-AR-ZT-09
Record Dates: First submitted 2024-05-06; First posted 2024-05-08 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Esophageal Achalasia
Keywords: Peroral Endoscopic Myotomy; anesthesia; Esophageal Achalasia
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild malnutrition: Patients will be divided into 3 groups according to the MUST malnutrition score in the preoperative period (BMI, weight loss, acute illness/oral feeding difficulty). (mild, moderate, severe malnutrition)
  Interventions: Other: MUST malnutrition score
- Moderate malnutrition: Patients will be divided into 3 groups according to the MUST malnutrition score in the preoperative period (BMI, weight loss, acute illness/oral feeding difficulty). (mild, moderate, severe malnutrition)
  Interventions: Other: MUST malnutrition score
- Severe malnutrition: Patients will be divided into 3 groups according to the MUST malnutrition score in the preoperative period (BMI, weight loss, acute illness/oral feeding difficulty). (mild, moderate, severe malnutrition)
  Interventions: Other: MUST malnutrition score

INTERVENTIONS:
Other: MUST malnutrition score — MUST malnutrition score

SUMMARY:
The hypothesis of this study is to investigate cardiorespiratory and renal complications in patients under general anesthesia undergoing POEM surgery.

DETAILED DESCRIPTION:
The primary purpose of this study is to define mild, medium and severe risk groups for malnutrition by using preoperative albumin values and MUST score in achalasia patients planned for POEM operation, and to determine the relationship of malnutrition/degree as well as demographic characteristics and comorbidities with postoperative respiratory and renal complications.

The secondary aim of this study was to determine persistent respiratory and renal outcome at 3 months after POEM procedure.

ELIGIBILITY:
Inclusion Criteria:

* Criteria for inclusion in the study:
* Patients diagnosed with achalasia and suitable for POEM treatment by gastroenterology physicians
* ASA 1-3
* Between the ages of 18-80

Exclusion Criteria:

* Criteria for exclusion from the study:
* Those with a known history of active lung infection, advanced COPD, or respiratory failure
* Patients with EF below 40%, severe ischemic heart failure, presence of valve disease
* Those with bleeding diathesis and severe thrombocytopenia (limit 30-50 thousand)
* severe kidney dysfunction
* In the presence of known intolerance or allergy to certain medications for sedation, analgesia, or both
* Pre-existing increased intracranial pressure
* Having a BMI >30
* Severe uncorrected hypovolemiaHistory of radiotherapy to the esophagus
* History of mucosal resection or ablation in the area where POEM will be applied
* Presence of cirrhosis and portal hypertension.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this retrospective cohort study, 50 patients diagnosed with achalasia who applied to the Gastroenterology department of Ümraniye Training and Research Hospital between October 2021 and February 2024 and were indicated for POEM treatment will be included.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
cardiorespiratory advers events | up to 12 weeks
  hypercapnia (above 45mmHg)
postoperative renal complications | up to 12 weeks
  serum creatinine 0.3 mg/dL rise

SECONDARY OUTCOMES:
Malnutrition condition | up to 12 weeks
  serum albumin (3.4 to 5.4 g/dL)
escart score | up to 12 weeks
  weight loss ( <5kg to10kg>)

CONTACTS AND LOCATIONS:
Locations (1):
- Umraniye Education and Research hospital, Istanbul, Turkey (Türkiye)